CLINICAL TRIAL: NCT00656136
Title: Phase IIb/III Randomized, Double-blind Trial of BIBW 2992 Plus Best Supportive Care (BSC) Versus Placebo Plus BSC in Non-small Cell Lung Cancer Patients Failing Erlotinib or Gefitinib (LUX-Lung 1)
Brief Title: BIBW 2992 and BSC Versus Placebo and BSC in Non-small Cell Lung Cancer Patients Failing Erlotinib or Gefitinib (LUX-LUNG 1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1200.23; 2007-005983-28 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Results first posted 2013-11-27 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

ARMS (2):
- Placebo (Placebo Comparator): Patients receive placebo once daily
  Interventions: Drug: placebo
- BIBW 2992 (Experimental): Patients receive BIBW 2992 tablets once daily
  Interventions: Drug: BIBW 2992

INTERVENTIONS:
Drug: placebo — Patients receive placebo once daily
  Arms: Placebo
Drug: BIBW 2992 — Patients receive afatinib tablets once daily, and can reduce dose for adverse event management. Afatinib is given once daily, continuously until disease progression or unacceptable toxicity.
  Arms: BIBW 2992

SUMMARY:
This randomized, double-blind, multi-center Phase IIb/III trial will be performed in patients with NSCLC who have received previous treatment with at least one but not more than two lines of cytotoxic chemotherapy (one line must have been a platinum-containing regimen) and either gefitinib or erlotinib for a period of at least 12 weeks and then progressed.

The primary objective of this randomized trial is to determine the efficacy of BIBW 2992 as a single agent (Arm A) as compared to a matching placebo (Arm B) in this patient population. Patients on both treatment arms will receive best supportive care in addition to study treatment.

Patients enrolled into the trial will be treated and followed until death or lost to follow-up.

ELIGIBILITY:
Inclusion criteria:

1. Patients with pathologic confirmation of NSCLC Stage III-B (with pleural effusion) or Stage IV adenocarcinoma who have failed at least one but not more than two lines of cytotoxic chemotherapy (including adjuvant chemotherapy). One of the chemotherapy regimens must have been platinum-based.
2. Progressive disease following at least 12 weeks of treatment with erlotinib (Tarceva®) or gefitinib (Iressa®)
3. Eastern Cooperative Oncology Group (ECOG, R01-0787) performance Score 0, 1 or 2
4. Patients with at least one tumor lesion that can accurately be measured by magnetic resonance imaging (MRI), or computed tomography (CT) in at least one dimension with longest diameter to be recorded as >20 mm using conventional techniques or >10 mm with spiral CT scan
5. Male and female patients age >18 years
6. Life expectancy of at least three (3) months
7. Written informed consent that is consistent with ICH-GCP guidelines

Exclusion criteria:

1. Use of erlotinib (Tarceva®) or gefitinib (Iressa®) within 14 days of treatment Day 1
2. Chemo-, hormone- (other than megestrol acetate or steroids required for maintenance non-cancer therapy) or immunotherapy within the past 4 weeks
3. Active brain metastases
4. Significant or recent acute gastrointestinal disorders with diarrhea
5. Patients who have any other life-threatening illness or organ system dysfunction,
6. Other malignancies diagnosed within the past five (5) years
7. Radiotherapy within the past 2 weeks prior to treatment
8. History of clinically significant or uncontrolled cardiac disease
9. Adequate ANC and platelet count
10. Adequate liver and kidney function
11. Patients with any serious active infection including known HIV, active hepatitis B or active hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 585 (Actual)
Dates: Start 2008-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (90):
- United States (14):
  - 1200.23.038 Boehringer Ingelheim Investigational Site, Kingman, Arizona
  - 1200.23.046 Boehringer Ingelheim Investigational Site, Fayetteville, Arkansas
  - 1200.23.027 Boehringer Ingelheim Investigational Site, Anaheim, California
  - 1200.23.028 Boehringer Ingelheim Investigational Site, Berkeley, California
  - 1200.23.029 Boehringer Ingelheim Investigational Site, Modesto, California
  - 1200.23.045 Boehringer Ingelheim Investigational Site, Montebello, California
  - 1200.23.009 Boehringer Ingelheim Investigational Site, Orange, California
  - 1200.23.026 Boehringer Ingelheim Investigational Site, Palm Springs, California
  - 1200.23.024 Boehringer Ingelheim Investigational Site, North Miami Beach, Florida
  - 1200.23.020 Boehringer Ingelheim Investigational Site, New York, New York
  - 1200.23.013 Boehringer Ingelheim Investigational Site, Valhalla, New York
  - 1200.23.056 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - 1200.23.039 Boehringer Ingelheim Investigational Site, Renton, Washington
  - 1200.23.050 Boehringer Ingelheim Investigational Site, Seattle, Washington
- Belgium (5):
  - 1200.23.32004 Boehringer Ingelheim Investigational Site, Edegem
  - 1200.23.32003 Boehringer Ingelheim Investigational Site, Ghent
  - 1200.23.32001 Boehringer Ingelheim Investigational Site, Leuven
  - 1200.23.32005 Boehringer Ingelheim Investigational Site, Liège
  - 1200.23.32006 Boehringer Ingelheim Investigational Site, Namur
- Canada (5):
  - 1200.23.1002 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1200.23.1005 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1200.23.1009 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1200.23.1001 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1200.23.1004 Boehringer Ingelheim Investigational Site, Montreal, Quebec
- China (9):
  - 1200.23.86001 Boehringer Ingelheim Investigational Site, Beijing
  - 1200.23.86002 Boehringer Ingelheim Investigational Site, Beijing
  - 1200.23.86003 Boehringer Ingelheim Investigational Site, Beijing
  - 1200.23.86009 Boehringer Ingelheim Investigational Site, Chengdu
  - 1200.23.86007 Boehringer Ingelheim Investigational Site, Guangzhou
  - 1200.23.86008 Boehringer Ingelheim Investigational Site, Hangzhou
  - 1200.23.86004 Boehringer Ingelheim Investigational Site, Shanghai
  - 1200.23.86005 Boehringer Ingelheim Investigational Site, Shanghai
  - 1200.23.86006 Boehringer Ingelheim Investigational Site, Shanghai
- France (11):
  - 1200.23.3303A Boehringer Ingelheim Investigational Site, Besançon
  - 1200.23.3303C Boehringer Ingelheim Investigational Site, Besançon
  - 1200.23.3305A Boehringer Ingelheim Investigational Site, Caen
  - 1200.23.3304A Boehringer Ingelheim Investigational Site, La Tronche
  - 1200.23.3304B Boehringer Ingelheim Investigational Site, La Tronche
  - 1200.23.3307A Boehringer Ingelheim Investigational Site, Lyon
  - 1200.23.3301A Boehringer Ingelheim Investigational Site, Paris
  - 1200.23.3302A Boehringer Ingelheim Investigational Site, Paris
  - 1200.23.3302B Boehringer Ingelheim Investigational Site, Paris
  - 1200.23.3306A Boehringer Ingelheim Investigational Site, Toulouse
  - 1200.23.3306C Boehringer Ingelheim Investigational Site, Toulouse
- Germany (8):
  - 1200.23.49010 Zentralklinik Bad Berka GmbH, Bad Berka
  - 1200.23.49002 Innere Klinik und Poliklinik (Tumorforschung), Essen
  - 1200.23.49003 Asklepios Fachkliniken München-Gauting, Gauting
  - 1200.23.49005 Krankenhaus Großhansdorf, Großhansdorf
  - 1200.23.49008 Universitätsklinik Hamburg-Eppendorf, Hamburg
  - 1200.23.49004 Johannes Gutenberg-Universität Mainz, Mainz
  - 1200.23.49001 Universitätsklinikum Mannheim, Mannheim
  - 1200.23.49006 HSK, Dr. Horst-Schmidt-Kliniken GmbH, Wiesbaden
- 1200.23.85202 Boehringer Ingelheim Investigational Site, Hong Kong, Hong Kong
- Italy (6):
  - 1200.23.39003 Boehringer Ingelheim Investigational Site, Genova
  - 1200.23.39007 Boehringer Ingelheim Investigational Site, Orbassano (TO)
  - 1200.23.39002 Boehringer Ingelheim Investigational Site, Perugia
  - 1200.23.39004 Boehringer Ingelheim Investigational Site, Prato
  - 1200.23.39008 Boehringer Ingelheim Investigational Site, Roma
  - 1200.23.39001 Boehringer Ingelheim Investigational Site, Rozzano (MI)
- Netherlands (3):
  - 1200.23.31002 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1200.23.31001 Boehringer Ingelheim Investigational Site, Groningen
  - 1200.23.31003 Boehringer Ingelheim Investigational Site, Helmond
- 1200.23.65001 Boehringer Ingelheim Investigational Site, Singapore, Singapore
- South Korea (6):
  - 1200.23.82005 Boehringer Ingelheim Investigational Site, Gyeonggi-do
  - 1200.23.82006 Boehringer Ingelheim Investigational Site, Hwasun
  - 1200.23.82001 Boehringer Ingelheim Investigational Site, Seoul
  - 1200.23.82002 Boehringer Ingelheim Investigational Site, Seoul
  - 1200.23.82003 Boehringer Ingelheim Investigational Site, Seoul
  - 1200.23.82004 Boehringer Ingelheim Investigational Site, Seoul
- Spain (6):
  - 1200.23.3405 Boehringer Ingelheim Investigational Site, Barcelona
  - 1200.23.3404 Boehringer Ingelheim Investigational Site, Cruces
  - 1200.23.3401 Boehringer Ingelheim Investigational Site, Madrid
  - 1200.23.3403 Boehringer Ingelheim Investigational Site, Madrid
  - 1200.23.3406 Boehringer Ingelheim Investigational Site, Madrid
  - 1200.23.3402 Boehringer Ingelheim Investigational Site, Valencia
- Taiwan (7):
  - 1200.23.88604 Taichung Veterans General Hospital, Taichung
  - 1200.23.88605 China Medical University Hospital, Taichung
  - 1200.23.88606 National Cheng Kung University Hospital, Tainan
  - 1200.23.88601 National Taiwan University Hospital, Taipei
  - 1200.23.88602 Veterans General Hospital, Taipei
  - 1200.23.88607 Tri-Service General Hospital, Taipei
  - 1200.23.88603 Chang Gung Memorial Hosp-Linkou, Taoyuan District
- Thailand (3):
  - 1200.23.66001 Boehringer Ingelheim Investigational Site, Chiang Mai
  - 1200.23.66003 Boehringer Ingelheim Investigational Site, Pathumwan, Bangkok
  - 1200.23.66002 Boehringer Ingelheim Investigational Site, Songkhla
- United Kingdom (5):
  - 1200.23.4404 Boehringer Ingelheim Investigational Site, Dundee
  - 1200.23.4403 Boehringer Ingelheim Investigational Site, Edinburgh
  - 1200.23.4401 Boehringer Ingelheim Investigational Site, Glasgow
  - 1200.23.4405 Boehringer Ingelheim Investigational Site, London
  - 1200.23.4406 Boehringer Ingelheim Investigational Site, Sutton

REFERENCES:
- [Derived] Miller VA, Hirsh V, Cadranel J, Chen YM, Park K, Kim SW, Zhou C, Su WC, Wang M, Sun Y, Heo DS, Crino L, Tan EH, Chao TY, Shahidi M, Cong XJ, Lorence RM, Yang JC. Afatinib versus placebo for patients with advanced, metastatic non-small-cell lung cancer after failure of erlotinib, gefitinib, or both, and one or two lines of chemotherapy (LUX-Lung 1): a phase 2b/3 randomised trial. Lancet Oncol. 2012 May;13(5):528-38. doi: 10.1016/S1470-2045(12)70087-6. Epub 2012 Mar 26. PMID 22452896

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two-arm, randomised (2:1 ratio), double-blind , placebo-controlled, multi-centre trial. 585 patients were randomised. All patients randomized received at least one dose of study medication.
Groups:
- Placebo Plus Best Supportive Care (BSC): Patients received matching placebo for 50 mg, 40 mg or 30 mg afatinib tablets starting with 50 mg/day. Dose reductions were managed in the same way as for the afatinib arm.
- Afatinib 50 mg/Day Plus Best Supportive Care (BSC): Patients started with a 50 mg/day dose. Dose reductions were permitted by the protocol to 40 mg/day plus Best Supportive Care (BSC) or 30 mg /day plus BSC based upon prespecified Adverse Events and Common Terminology Criteria for Adverse Events (CTCAE) grade (Version 3.0).
Period: Overall Study
Arm/Group | Placebo Plus Best Supportive Care (BSC) | Afatinib 50 mg/Day Plus Best Supportive Care (BSC)
Started | 195 (Randomised patients.) | 390 (Randomised patients.)
Completed | 0 | 0
Not Completed | 195 | 390
Not completed — Progressive disease | 177 | 322
Not completed — Other Adverse Event | 5 | 51
Not completed — Protocol Violation | 2 | 3
Not completed — Patient refused to take study medication | 7 | 10
Not completed — Unknown and others | 4 | 4

BASELINE CHARACTERISTICS:
Population: Randomized Set (RS) included all patients randomised to receive treatment
Groups:
- Afatinib 50 mg/Day Plus Best Supportive Care (BSC): Patients started with a 50 mg/day dose. Dose reductions were permitted by the protocol to 40 mg/day plus BSC or 30 mg /day plus BSC based upon prespecified Adverse Events and Common Terminology Criteria for Adverse Events (CTCAE) grade (Version 3.0).
- Total: Total of all reporting groups
Arm/Group | Placebo Plus Best Supportive Care (BSC) | Afatinib 50 mg/Day Plus Best Supportive Care (BSC) | Total
Number analyzed (Participants) | 195 | 390 | 585
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (10.4) | 58 (10.8) | 58 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 231 | 348
  Male | 78 | 159 | 237
Race/Ethnicity, Customized [Number; unit: Number of participants]
  Caucasian | 72 | 121 | 193
  Eastern Asian | 110 | 227 | 337
  Other Asian | 12 | 38 | 50
  Other | 1 | 4 | 5
Baseline Eastern Cooperative Oncology Group (ECOG) performance score [Number; unit: Number of participants] — ECOG Performance Score was measured on 6 point scale where 0="Fully active", 1="Restricted in physically strenuous activity" and 2="Ambulatory and capable of all self care but unable to carry out any work activities", 3="Capable of only limited self care, confined to bed or chair 50% or more of waking hours", 4="Bedbound", and 5="Death".
  Number of participants
    ECOG score = 0 | 53 | 92 | 145
    ECOG score = 1 | 127 | 268 | 395
    ECOG score = 2 | 15 | 30 | 45

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was the duration from the date of randomization to the date of death. Patients who were alive were censored at the last contact date prior to the database lock.
  For the primary analysis 11 patients were lost to follow-up and were censored at the last contact date when they were known to be still alive. Primary analysis data cut-off date was 08 July 2010.
  For the final analysis 13 patients were lost to follow-up and were censored at the last contact date when they were known to be still alive. Final analysis data cut-off date was 04 October 2013.
Time Frame: From randomization until death or the last patient out date, an average of 12 months
Population: Randomized set was all patients who were randomized and for this study all of these patients received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo Plus Best Supportive Care (BSC) | Afatinib 50 mg/Day Plus Best Supportive Care (BSC)
Number analyzed (Participants) | 195 | 390
Months
  Primary analysis (358 deaths) | 11.96 [10.15 to 14.26] | 10.78 [9.95 to 11.99]
  Final analysis (526 deaths) | 11.73 [10.05 to 14.06] | 10.87 [9.95 to 12.25]
Statistical Analysis 1: Comparison: Placebo Plus Best Supportive Care (BSC) vs Afatinib 50 mg/Day Plus Best Supportive Care (BSC); Primary analysis was performed after 358 deaths were observed among randomized patients. The data cut-off date for the primary analysis was 08 July 2010; Test type: Superiority or Other; p = 0.7428, Regression, Cox — P-value is one-sided (afatinib vs placebo) log rank test stratified by gender and baseline ECOG score (0,1 vs 2); Model stratified by gender and baseline ECOG score (0,1 vs 2); Hazard Ratio (HR) = 1.077, 95% CI 2-sided [0.862 to 1.346]
Statistical Analysis 2: Comparison: Placebo Plus Best Supportive Care (BSC) vs Afatinib 50 mg/Day Plus Best Supportive Care (BSC); Final analysis was performed after 526 deaths were observed among randomized patients. The data cut-off date for the final analysis was 04 October 2013; Test type: Superiority or Other; p = 0.3955, Regression, Cox — P-value is one-sided (afatinib vs placebo) log rank test stratified by gender and baseline ECOG score (0,1 vs 2); Model stratified by gender and baseline ECOG score (0,1 vs 2); Hazard Ratio (HR) = 0.976, 95% CI 2-sided [0.814 to 1.170]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as time from randomisation to disease progression or death whichever occurs first. Assessed by central independent review according to the Response Evaluation Criteria in Solid Tumours version 1.0 (RECIST 1.0).
Time Frame: From randomization to disease progression, death or the data cutoff on 07 July 2010, an average of 3.3 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo Plus Best Supportive Care (BSC) | Afatinib 50 mg/Day Plus Best Supportive Care (BSC)
Number analyzed (Participants) | 195 | 390
Months | 1.08 [0.95 to 1.68] | 3.29 [2.79 to 4.40]
Statistical Analysis 1: Comparison: Placebo Plus Best Supportive Care (BSC) vs Afatinib 50 mg/Day Plus Best Supportive Care (BSC); Test type: Superiority or Other; p < 0.0001, Regression, Cox — P-value is one-sided (afatinib vs placebo) log rank test stratified by gender and baseline ECOG score (0,1 vs 2); Model stratified by gender and baseline ECOG score (0,1 vs 2); Hazard Ratio (HR) = 0.381, 95% CI 2-sided [0.306 to 0.475]

3. Secondary Outcome: Objective Response Rate (OR)
Description: OR is defined as complete response (CR) and partial response (PR). Assessed by central independent review according to RECIST 1.0.
Time Frame: From randomization to disease progression, death or the data cutoff on 07 July 2010, an average of 3.3 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of patients with OR
Arm/Group | Placebo Plus Best Supportive Care (BSC) | Afatinib 50 mg/Day Plus Best Supportive Care (BSC)
Number analyzed (Participants) | 195 | 390
Percentage of patients with OR | 0.5 [0.0 to 2.8] | 7.4 [5.0 to 10.5]
Statistical Analysis 1: Comparison: Placebo Plus Best Supportive Care (BSC) vs Afatinib 50 mg/Day Plus Best Supportive Care (BSC); Test type: Superiority or Other; p = 0.0071, Regression, Logistic — P-value is derived from logistic regression model adjusted for stratification factors, gender and baseline ECOG score (0, 1 vs 2); Model stratified by gender and baseline ECOG score (0,1 vs 2); Odds Ratio (OR) = 15.61, 95% CI 2-sided [2.1 to 115]

ADVERSE EVENTS:
Time Frame: From the date of first drug intake up to 28 days after the last drug intake for on-treatment adverse events or the last patient out date on 4 October 2013.
Groups:
- Placebo: Patients received matching placebo for 50 mg, 40 mg or 30 mg afatinib tablets starting with 50 mg/day. Dose reductions were managed in the same way as for the afatinib arm.
- Afatinib 50 mg/Day: Patients started with a 50 mg/day dose. Dose reductions were permitted by the protocol to 40 mg/day plus BSC or 30 mg /day plus BSC based upon prespecified Adverse Events and Common Terminology Criteria for Adverse Events (CTCAE) grade (Version 3.0).
Arm/Group | Placebo | Afatinib 50 mg/Day
Serious Adverse Events (participants affected / at risk) | 36/195 | 136/390
Other Adverse Events (participants affected / at risk) | 167/195 | 383/390
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=195) | Afatinib 50 mg/Day (N=390)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 2
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 2
Sick sinus syndrome (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Blindness (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Eye movement disorder (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 18
Dysphagia (Gastrointestinal disorders) | 3 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 4
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 4
Proctalgia (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 1 | 5
Asthenia (General disorders) | 1 | 1
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 2 | 0
Condition aggravated (General disorders) | 0 | 1
Death (General disorders) | 1 | 3
Extravasation (General disorders) | 0 | 1
Face oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 3
General physical health deterioration (General disorders) | 1 | 2
Hernia (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Medical device complication (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 2
Pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 7
Sudden cardiac death (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Atypical pneumonia (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Candida infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Lower respiratory tract infection fungal (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 4
Paronychia (Infections and infestations) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 10
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 5
Soft tissue infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 4
Blood culture positive (Investigations) | 0 | 1
Blood potassium increased (Investigations) | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 1
Prostatic specific antigen increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 16
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 11
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1
Brain mass (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 2
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Convulsion (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 3
Dysarthria (Nervous system disorders) | 1 | 0
Embolic cerebral infarction (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 2
Ischaemic stroke (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Paraplegia (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 2
Tremor (Nervous system disorders) | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 1 | 1
Delirium (Psychiatric disorders) | 0 | 1
Acute prerenal failure (Renal and urinary disorders) | 0 | 1
Oliguria (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 7
Renal impairment (Renal and urinary disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 14
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 9
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 5
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 2
Thrombosis (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=195) | Afatinib 50 mg/Day (N=390)
Anaemia (Blood and lymphatic system disorders) | 3 | 23
Abdominal pain upper (Gastrointestinal disorders) | 8 | 25
Constipation (Gastrointestinal disorders) | 24 | 43
Diarrhoea (Gastrointestinal disorders) | 18 | 334
Mouth ulceration (Gastrointestinal disorders) | 0 | 51
Nausea (Gastrointestinal disorders) | 39 | 90
Stomatitis (Gastrointestinal disorders) | 2 | 82
Vomiting (Gastrointestinal disorders) | 25 | 75
Asthenia (General disorders) | 16 | 36
Chest pain (General disorders) | 11 | 27
Fatigue (General disorders) | 23 | 72
Mucosal inflammation (General disorders) | 2 | 95
Pyrexia (General disorders) | 7 | 36
Folliculitis (Infections and infestations) | 0 | 25
Paronychia (Infections and infestations) | 1 | 131
Weight decreased (Investigations) | 2 | 37
Decreased appetite (Metabolism and nutrition disorders) | 22 | 118
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 29
Back pain (Musculoskeletal and connective tissue disorders) | 22 | 29
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 20
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 27
Dizziness (Nervous system disorders) | 6 | 20
Dysgeusia (Nervous system disorders) | 1 | 22
Headache (Nervous system disorders) | 9 | 21
Insomnia (Psychiatric disorders) | 10 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 36 | 54
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 54
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 73
Productive cough (Respiratory, thoracic and mediastinal disorders) | 13 | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 42
Acne (Skin and subcutaneous tissue disorders) | 0 | 27
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 28
Dry skin (Skin and subcutaneous tissue disorders) | 14 | 62
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 30
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 73
Rash (Skin and subcutaneous tissue disorders) | 23 | 248
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.